CLINICAL TRIAL: NCT04153617
Title: Nutritional and Clinical Trial to Evaluate the Effect of a Modified Honey With Soluble Fiber and Polyphenols Consumption in Subjects With Overweight/Obesity and Dyslipidemia
Brief Title: Enriched Honey With Soluble Fiber and Polyphenols on Satiety and Dyslipidemia
Acronym: SACIMIEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Primo Mendoza S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HULP 5049
Record Dates: First submitted 2019-09-12; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-09

CONDITIONS: Overweight and Obesity; Dyslipidemias
Keywords: Saciety; Honey; Fiber; Polyphenols; Visual Analogue Scale; Cross-over; Parallel
MeSH Terms: conditions — Overweight; Obesity; Dyslipidemias | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control honey (Placebo Comparator): Orange blossom honey.
  Middle term trial: 40g/day for 3 months in two daily intakes of 20 g/day.
  Short term trial: 20g/day in a single day.
  Interventions: Dietary Supplement: Control honey; Dietary Supplement: Modified honey with soluble fiber and polyphenols
- Modified honey with soluble fiber and polyphenols (Experimental): Honey modified with soluble fiber and polyphenols
  Middle term trial: 40g/day for 3 months in two daily intakes of 20 g/day.
  Short term trial: 20g/day in a single day.
  Interventions: Dietary Supplement: Control honey; Dietary Supplement: Modified honey with soluble fiber and polyphenols

INTERVENTIONS:
Dietary Supplement: Control honey — Control honey defined as orange blossom honey. Intake daily for 3 months (40 g/day)
Dietary Supplement: Modified honey with soluble fiber and polyphenols — Honey modified with soluble fiber and polyphenols, with same organoleptic conditions as control honey. Intake daily for 3 months (40 g/day)

SUMMARY:
The aim of this trial is to evaluate the possible benefits on saciety and dyslipidemia in subjects with overweight/obesity (BMI ≥25 y <40 kg / m2) and dyslipemia after consumption of a modifed honey with soluble fiber and polyphenols.

Some studies have shown the contribution of high-fiber foods in the reduction of the cardiovascular risk. Besides, polyphenols have reported with their potent antioxidant effect and their implication lowering the vardiovascular risk.

DETAILED DESCRIPTION:
The trial was designed as a randomized, parallel, double-blind and controlled study with 2 experimental arms. This study was performed to evaluate the effect on saciety and dyslipidemia of subjects with overweight/obesity after a long consumption (3 months) of a modified honey with soluble fiber and polyphenols. Additionally, a short-term randomized, cross-over, doble-blind and controlled trial was also performed to evaluate immediate saciety effect on the same subjects.

For the middle-term study, investigators included 67 participants (8 men and 59 women) between 18 and 65 years (BMI ≥25 and <40 kg / m2). All volunteers were randomized into 2 study groups, and participants received the 2 different study products during the 3 months. On the other hand, the associated short-term trial included 10 participants (5 men and 5 women) between 18 and 65 years (BMI ≥25 and <40 kg / m2). All volunteers were randomized into 2 study groups, and participants took the 2 different study products in two non-consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years old.
* Body Mass Index (BMI) ≥25 and <40 kg/m2.
* Cardiovascular risk <10% to 10 years measured by REGICOR.
* Total cholesterol ≥ 200 mg/d and at least 2 factors included in the following list:

  * ≥ 45 years or women ≥ 55 years.
  * Family history of cardiovascular disease (CVD) in first degree male relative less than 55 years of age and less than 65 years in women.
  * HDL cholesterol: men <40 or women <50.
  * Triglycerides ≥ 150mg/dL and <200 mg/dL
  * LDL cholesterol ≥ 130mg/dL and < 160mg/dL
  * Smoker
* Willingness to follow a healthy and balanced hypocaloric diet with mandatory physical activity
* Social or familiar environment that prevents from accomplishing the dietary treatment
* Adequate cultural level and understanding for the clinical trial.
* Signed informed consent

Exclusion Criteria:

* Body Mass Index (BMI) <25 and ≥40 kg/m2.
* Individuals diagnosed with Diabetes Mellitus type 1 or 2.
* Individuals with dyslipidemia on pharmacological treatment.
* Individuals with hypertension on pharmacological treatment.
* Individuals diagnosed with eating disorders.
* Individuals fructose-intolerant.
* Individuals with a diagnosis of celiac disease or a gluten intolerance.
* Individuals with severe chronic diseases (hepatic, kidney, …)
* Individuals receiving a pharmacological treatment that modifies the lipid or glucose profile.
* Individuals who have participated in the last 3 months in a program or clinical trial to lose weight.
* Individuals with mental illness.
* Smokers wanting to stop to smoke during the period that clinical trial lasts.
* Individuals with high alcohol consumption (> 2-3 servings/ day in men and> 1 serving/day in women (1 serving = 1 glass of wine or 1 bottle of beer).
* Individuals with large weight fluctuations of more than 4 kg or who have undergone in six months a weight loss diet.
* Individuals with sensory problems.
* Individuals with gastrointestinal diseases that affect the digestion or absorption of nutrients.
* Individuals under pharmacological treatment for losing weight unless treatment is suspended 30 days before the start of the trial.
* Subjects with intense physical activity.
* Subjects with food allergies to meals included in breakfast, study product or lunch or that reject their consumption
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Satiety Hunger Assessment | Day 1, 2
  Visual Analogue Scale (VAS). 100mm horizontal line anchored at each end with the extremes of the subjective feeling to be quantified. Subjects are instructed to rate the sensation being experienced according to how they define the line.
  e.g., "not at all hungry" (0mm) and "as hungry as I have ever felt" (100mm). Multiple measures are taken at repeated time intervals described below.

SECONDARY OUTCOMES:
Change from Baseline Lipid Metabolism Parameters | Week 1,12
  Cholesterol, LDL-C, HDL-C, TG
Amount of food consumed in a "food ad libitum" | Day 1, 2
  120 min After eating the study product
Total amount of food consumed in 24h | Day 1, 2; Week 1, 6, 12
  24h Food Record Method
Change from Baseline Glucose Metabolism Parameters | Day 1, 2; Week 1, 12
  Glucose
Anthropometric Parameters | Day 1, 2; Week 1, 12
  Weight and height will be combined to report BMI in kg/m2
Sensory Perception Test | Day 1, 2; Week 6, 12
  Questionnaire of analysis of sensory perception of the food study product. Five questions that are valued on a scale of 0% to 100% asking about the taste and smell of the study product: desire with which the product is taken, taste, smell, consistency and what wait for effectiveness.
Adverse Effects | Day 1, 2; Week 6, 12
  Gastrointestinal Symptoms (Nausea, Diarrhea, Bloating and other disorders)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, MD, Phd, Principal Investigator — La Paz University Hospital
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No